CLINICAL TRIAL: NCT03915119
Title: Genetic Fuzzy Artificial Intelligence Driven Virtual Reality for Prevention of Collision-based Injury
Brief Title: Fuzzy AI Using VR for Collision Prevention
Acronym: CAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2017-6006
Record Dates: First submitted 2018-10-30; First posted 2019-04-16 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Injuries
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR Obstacle group (Experimental): Initial Visit: navigates a cluttered array of fixed and moving virtual obstacles to reach a way-point (goal) as fast and efficiently (avoiding obstacles) as possible. In each block, task difficulty (i.e., complexity) will increase linearly, regardless of success or failure (≥ 1 collision before reaching the goal).
  Second (Training) Visit (randomized into two groups):
  Interventions: Other: GFT AI training
- Agility Group (Experimental): Initial Visit: Completes a soccer ball dribbling agility task in which they must dribble a soccer ball toward an artificial way-point, while avoiding artificial obstacles overlaid onto the real world via a Microsoft Hololens augmented reality display.
  Second (Training) Visit
  Interventions: Other: GFT AI training

INTERVENTIONS:
Other: GFT AI training — navigates a cluttered environment of stationary and moving/pursuing virtual obstacles to reach a way-point as quickly and efficiently as possible. Block order and difficulty, as well as the behavior of the obstacles in each block, will be driven by the AI and statistically weighted to specifically target the perceptual-motor and neuromechanical mechanisms based on each athlete's visit 1 performance

SUMMARY:
The purpose of this study is to develop and test a VR training system that integrates GFT AI with virtual obstacle scenarios that, when compared to a sham-VR training system, is hypothesized to increase neuromechanical and perceptual-motor fitness, decrease collision frequency and impact forces for soccer athletes, during a single training session and also when assessed at approximately 1 week and 1 month following training.

DETAILED DESCRIPTION:
Player collisions cause over 70% of concussion injuries in contact sports, in addition to 50% of lower extremity injuries and 40% of catastrophic knee ligament injuries. The majority of these collisions are unanticipated, and associated with reduced neuromechanical and perceptual-motor fitness underlying an athlete's adaptability to on-field conditions. Thus, training collision anticipation necessitates a method that taps into neuromechanical and perceptual-motor fitness. Virtual reality (VR) is a tool that can target these mechanisms, while providing a safe, well-controlled environment for assessment and training. The current proposal innovates on VR with the integration of genetic fuzzy tree (GFT) artificial intelligence (AI) to drive scenario configuration designed to target modifiable mechanisms and tailored to the individual athlete's performance capabilities, for the optimization of behavior modification and skill transfer. The current study will examine test a GFT AI-driven VR collision anticipation training compared to a sham-VR training system in healthy soccer athletes.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* varsity high school or collegiate soccer athlete

Exclusion Criteria:

* unable to participate in soccer
* history of congenital or acquired cognitive, ophthalmologic, or neurological disorders including developmental delay, brain tumor, stroke, or known peripheral or central vestibular disorders
* patients who have begun anti-depressant, stimulant or anti-seizure medications for treatment of their symptoms or for other, unrelated reasons within two months of testing will be excluded from testing

Ages: 14 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Pro-saccades test | 10 minutes
  Pro-saccades will be tested as participants track discrete target motion that will jump randomly by 14, 16, 18, 20, 22, or 24˚ on the screen in a horizontal and vertical direction, at intervals varying pseudo randomly between 1.0 and 2.0 s. The current fixation target will be extinguished at the same time as the next peripheral target appears. The test sequence will take 30 s/trial (2 trials) and all participants will be instructed to follow the targets as quickly and accurately as possible

SECONDARY OUTCOMES:
Self paced saccades | 10 minutes
  Self-paced saccades will be assessed as the participant glances back and forth as quickly and accurately as possible between two constantly visual targets at ± 15˚ horizontally from one another. This test will take 30 s per trial and the participant will perform 2 trials.
Anti-saccades test | 10 minutes
  Anti-saccades will be tested as participants are presented discrete targets that jump randomly by 14, 16, 18, 20, 22, or 24˚ on the screen in a horizontal and vertical direction, at intervals varying pseudo randomly between 1.0 and 2.0 s while a cross-hairs is present in the center of the screen. The athletes will be instructed to fixate on the cross-hairs and at the moment each object appears, to saccade in the opposite direction and then return their gaze back to the cross-hairs for the start of the next trial.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Kiefer, PhD, Principal Investigator — Cincinanti Childrens Hospital
Locations (1):
- Cincinanti Childrens Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No